CLINICAL TRIAL: NCT02340598
Title: Prospective Randomized Pilot Study of the Effects of Cold Vests on Cardiovascular Risk Markers and Basal Metabolic Rate
Brief Title: Pilot Study of Effects of Cold Vests on Cardiovascular Risk Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Fredrik H Nystrom, Professor, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014/432-31
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Cardiovascular Risk Factors; Basal Metabolic Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cold vest (Experimental): Participants are given a cold vest that the pre-cool in a freezer. They are encouraged to use it daily to activate metabolism through brown adipose tissue and shivering.
  Interventions: Other: cold vest
- control (No Intervention): No intervention, just recording of risk factors and basal metabolic rate.

INTERVENTIONS:
Other: cold vest — The lowering of body temperature increases basal metabolic rate
  Arms: cold vest

SUMMARY:
Randomized trial of supplying a cold vest as compared with controls (no cold vest) on cardiovascular risk factors such as blood lipids, insulin, blood pressure and body weight and also on basal metabolic rate. Recruitment of 100 participants and 70 are randomized to being given a vest which they can use to increase basal metabolic rate during 1-2 hours (as long as the pre-cooled vest stays cool) by activating brown adipose tissue and/or shivering. The remaining 30 subjects will constitute a control group. Lab tests and anthropometrics are checked at baseline, after 2 months and after 1 year.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects that have no known metabolic relevant diseases

Exclusion Criteria:

* thyroid disease,
* mental disorders,
* language problems

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
basal metabolic rate | up to 1 year
  basal metabolic rate measured in the fasting state by indirect calorimetry
Composite measure of cardiovascular risk factors | up to 1 year
  Blood lipids, insulin, body weight, blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik H Nystrom, professor, Principal Investigator — Linkoeping University
Locations (1):
- University Hospital of Linkoping, Linköping, Sweden